CLINICAL TRIAL: NCT03031847
Title: Cardiac Resynchronization in the Elderly: Piloting Pacemaker vs. Defibrillator Therapy (Randomized Trial)
Brief Title: Cardiac Resynchronization in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samir Saba (Other)
Responsible Party: Sponsor-Investigator, Samir Saba, Associate Professor; Associate Chief of Cardiology; Director of Cardiovascular Electrophysiology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO17010015
Record Dates: First submitted 2017-01-19; First posted 2017-01-26 (Estimated); Results first posted 2022-08-23 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, controlled trial of CRT-P vs. CRT-D in HF patients (age ≥ 75 years)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Randomized- Pacemaker (CRT-P) (Other): Cardiac resynchronization therapy Pacemaker
  Interventions: Device: Cardiac Resynchronization Therapy Pacemaker
- Randomized- Defibrillator (CRT-D) (Other): Cardiac resynchronization therapy Defibrillator
  Interventions: Device: Cardiac Resynchronization Therapy Defibrillator
- Observational- Pacemaker (CRT-P) (Other): Cardiac resynchronization therapy Pacemaker (CRT-P): Patients in this arm declined randomization in the trial and elected to participate in the observational registry
  Interventions: Device: Cardiac Resynchronization Therapy Pacemaker
- Observational- Defibrillator (CRT-D) (Other): Cardiac resynchronization therapy Defibrillator (CRT-D): Patients in this arm declined randomization in the trial and elected to participate in the observational registry
  Interventions: Device: Cardiac Resynchronization Therapy Defibrillator

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy Pacemaker — Patients randomized to the pacemaker arm will receive a CRT-P device.
  Other Names: CRT-P
  Arms: Observational- Pacemaker (CRT-P); Randomized- Pacemaker (CRT-P)
Device: Cardiac Resynchronization Therapy Defibrillator — Patients randomized to the defibrillator arm will receive a CRT-D device.
  Other Names: CRT-D
  Arms: Observational- Defibrillator (CRT-D); Randomized- Defibrillator (CRT-D)

SUMMARY:
This pilot will enroll 50 HF patients (age ≥ 75 years) undergoing CRT device implantation at the hospitals of the University of Pittsburgh Medical Center, Duke University, Ohio State University, and the VA Pittsburgh Healthcare System. Patients will be randomized to CRT-P versus CRT-D and followed until study end. Rates of patient screening, enrollment, randomization, and retention as well as cost of care will be examined. The results of this pilot study will inform the design of a large pivotal non-inferiority trial and will be necessary for its success. Patients who refuse participation in the randomized pilot trial will be asked to enroll in a prospective observational cohort. Characteristics of patients who choose CRT-P vs. CRT-D will be compared and patients' level of satisfaction with their device decision will be measured.

DETAILED DESCRIPTION:
The goal of this study is to pilot test a randomized, controlled, non-inferiority trial comparing the survival and quality of life (QOL) of older patients receiving cardiac resynchronization therapy (CRT) pacemaker (CRT-P) versus defibrillator (CRT-D) therapy. This pilot will enroll 50 HF patients (age ≥ 75 years) undergoing CRT device implantation at the hospitals of the University of Pittsburgh Medical Center, Duke University, Ohio State University, and the VA Pittsburgh Healthcare System. Patients will be randomized to CRT-P versus CRT-D and followed until study end. Rates of patient screening, enrollment, randomization, and retention as well as cost of care will be examined. The results of this pilot study will inform the design of a large pivotal non-inferiority trial and will be necessary for its success. Patients who refuse participation in the randomized pilot trial will be enrolled and followed as part of a prospective observational cohort. Characteristics of patients who choose CRT-P vs. CRT-D will be compared and patients' level of satisfaction with their device decision will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 75 years
2. Left Ventricular Ejection Fraction (LVEF) ≤ 35% by cardiac imaging including echocardiogram, nuclear imaging, cardiac catheterization, or cardiac magnetic resonance imaging
3. QRS width >120 ms on surface electrocardiogram
4. New York Heart Association class II, III, or ambulatory IV for Heart Failure (HF)
5. Patient undergoing de novo CRT device implantation of CRT-D device change-out for battery depletion

Exclusion Criteria:

1. Patient within 40 days of acute myocardial infarction
2. Patient within 3 months of cardiac revascularization (percutaneous coronary intervention or bypass surgery)
3. Patient with prior history of cardiac arrest or documented sustained ventricular arrhythmia
4. Patient with expected longevity < 1 year
5. Patient not on optimal medical therapy for HF management including when tolerated β-blockers, angiotensin converting enzyme inhibitors or angiotensin receptor blockers
6. Patient not planning to have his/her follow-up at participating institution
7. Patient unable or unwilling to sign a written informed consent
8. Patient's with dementia that are unable to consent for themselves
9. Participating in any other clinical trials (observational/registries allowed)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Saba, MD, Principal Investigator — University of Pittsburgh
Locations (6):
- United States (6):
  - Duke University Health System, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - UPMC Hamot, Erie, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Veterans Research Foundation of Pittsburgh, Pittsburgh, Pennsylvania
  - UPMC Pinnacle, Wormleysburg, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dhande M, Myaskovsky L, Althouse A, Singh M, Weiss R, Shalaby A, Al-Khatib SM, Topoll A, Jain S, Saba S. Quality of Life and Type of Cardiac Resynchronization Therapy Device in Older Heart Failure Patients. J Palliat Med. 2023 Apr;26(4):481-488. doi: 10.1089/jpm.2022.0217. Epub 2022 Nov 8. PMID 36350362
- [Derived] Althouse AD, Jain SK, Shalaby A, Singh M, Weiss R, Myaskovsky L, Al-Khatib SM, Saba S. Feasibility of a Randomized Clinical Trial of Cardiac Resynchronization Therapy With or Without an Implantable Defibrillator in Older Patients. Circ Arrhythm Electrophysiol. 2022 Apr;15(4):e010795. doi: 10.1161/CIRCEP.121.010795. Epub 2022 Mar 31. No abstract available. PMID 35357219

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized- Pacemaker (CRT-P): Patients assigned to the pacemaker arm will receive CRT-P device
- Randomized- Defibrillator (CRT-D): Patients assigned to the defibrillator arm will receive CRT-D device
- Observational- Pacemaker (CRT-P): Patients in observational arm that chose CRT-P device
- Observational- Defibrillator (CRT-D): Patients in observational arm that chose CRT-D device
Period: Overall Study
Arm/Group | Randomized- Pacemaker (CRT-P) | Randomized- Defibrillator (CRT-D) | Observational- Pacemaker (CRT-P) | Observational- Defibrillator (CRT-D)
Started | 22 | 20 | 18 | 42
Completed | 20 | 18 | 14 | 36
Not Completed | 2 | 2 | 4 | 6
Not completed — Death | 1 | 1 | 2 | 3
Not completed — Lost to Follow-up | 1 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized- Pacemaker (CRT-P) | Randomized- Defibrillator (CRT-D) | Observational- Pacemaker (CRT-P) | Observational- Defibrillator (CRT-D) | Total
Number analyzed (Participants) | 22 | 20 | 18 | 42 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 22 | 20 | 18 | 42 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.7 (4.3) | 81.4 (4.9) | 84.7 (4.6) | 80.6 (4.0) | 81.5 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 6 | 8 | 28
  Male | 15 | 13 | 12 | 34 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 21 | 20 | 18 | 42 | 101
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 3 | 5
  White | 20 | 18 | 18 | 38 | 94
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 22 | 20 | 18 | 42 | 102

OUTCOME MEASURES:

1. Primary Outcome: Enrollment
Description: Rates of enrollment of participants in this randomized trial
Time Frame: At 1 year after start of the study
Population: Participants Enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized- Pacemaker (CRT-P) | Randomized- Defibrillator (CRT-D) | Observational- Pacemaker (CRT-P) | Observational- Defibrillator (CRT-D)
Number analyzed (Participants) | 22 | 20 | 18 | 42
Participants | 22 | 20 | 18 | 42

2. Secondary Outcome: QOL
Description: Quality of life of CRT-P versus CRT-D recipients using Minnesota Living with Heart Failure Questionnaires. The Minnesota Living with Heart Failure scale ranges from 0 to 105, in which a lower score indicates a better outcome. The Minnesota Living with Heart Failure Physical subscale ranges from 0 to 40 and the Minnesota Living with Heart Failure Mental subscale ranges from 0 to 25. Lower scores on the subscales indicate a better outcome.
Time Frame: At 6 months after enrollment
Population: Only participants with complete 6-month data for QoL assessments were reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized- Pacemaker (CRT-P) | Randomized- Defibrillator (CRT-D) | Observational- Pacemaker (CRT-P) | Observational- Defibrillator (CRT-D)
Number analyzed (Participants) | 17 | 17 | 12 | 32
score on a scale
  Overall QOL: MLWHF Questionnaire | 31.5 (30.3) | 16.1 (19.6) | 18.4 (9.6) | 37.8 (24.3)
  Physical QOL | 14.1 (13.8) | 8.2 (9.4) | 10.7 (7.7) | 18.9 (11.2)
  Emotional QOL | 7.0 (7.9) | 3.5 (5.4) | 2.9 (2.8) | 7.5 (7.0)

3. Secondary Outcome: QOL2
Description: QOL of CRT-P versus CRT-D recipients using RAND-36. The RAND-36 is a normalized scale with a range of 0 to 100, in which a higher score is indicative of a better outcome. PCS-T and MCS-T are the two summary components of the RAND-36. The subscales PCS-T and MCS-T are both normalized with a range of 0 to 100. Higher scores on the subscales indicate a better outcome.
Time Frame: At 6 months after enrollment
Population: Only participants with complete 6-month data for QoL assessments were reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized- Pacemaker (CRT-P) | Randomized- Defibrillator (CRT-D) | Observational- Pacemaker (CRT-P) | Observational- Defibrillator (CRT-D)
Number analyzed (Participants) | 17 | 17 | 12 | 32
score on a scale
  Rand-36: PCS-T | 37.4 (14.5) | 45.0 (12.4) | 37.7 (10.5) | 35.0 (11.2)
  Rand-36: MCS-T | 49.0 (13.4) | 51.4 (10.4) | 51.6 (10.4) | 47.7 (13.7)

4. Secondary Outcome: Retention
Description: Rates of retention of participants in this randomized trial
Time Frame: At 6 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized- Pacemaker (CRT-P) | Randomized- Defibrillator (CRT-D) | Observational- Pacemaker (CRT-P) | Observational- Defibrillator (CRT-D)
Number analyzed (Participants) | 22 | 20 | 18 | 42
Participants | 17 | 17 | 12 | 32

5. Secondary Outcome: Health Care Cost
Description: Cost of health care between CRT-P and CRT-D recipients.
Time Frame: At 6 months after enrollment
Population: Data was not collected
Arm/Group | Randomized- Pacemaker (CRT-P) | Randomized- Defibrillator (CRT-D) | Observational- Pacemaker (CRT-P) | Observational- Defibrillator (CRT-D)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 months.
Description: Adverse events were collected and classified as serious or not serious, cardiac or not cardiac. Cardiac events were further differentiated by arrhythmic or non-arrhythmic. Adverse events were not classified by specific organ system.
Arm/Group | Randomized- Pacemaker (CRT-P) | Randomized- Defibrillator (CRT-D) | Observational- Pacemaker (CRT-P) | Observational- Defibrillator (CRT-D)
All-Cause Mortality (participants affected / at risk) | 3/22 | 3/20 | 6/18 | 17/42
Serious Adverse Events (participants affected / at risk) | 6/22 | 3/20 | 9/18 | 18/42
Other Adverse Events (participants affected / at risk) | 9/22 | 6/20 | 2/18 | 13/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized- Pacemaker (CRT-P) (N=22) | Randomized- Defibrillator (CRT-D) (N=20) | Observational- Pacemaker (CRT-P) (N=18) | Observational- Defibrillator (CRT-D) (N=42)
Cardiac (Cardiac disorders) | 2 | 1 | 4 | 14
Non-Cardiac (General disorders) | 4 | 3 | 7 | 7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized- Pacemaker (CRT-P) (N=22) | Randomized- Defibrillator (CRT-D) (N=20) | Observational- Pacemaker (CRT-P) (N=18) | Observational- Defibrillator (CRT-D) (N=42)
Cardiac (Cardiac disorders) | 5 | 3 | 0 | 9
Non-Cardiac (General disorders) | 6 | 4 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/47/NCT03031847/Prot_SAP_000.pdf